CLINICAL TRIAL: NCT00546247
Title: A Phase 1/2, Ascending Multiple-Dose Study to Evaluate the Safety, Efficacy and Pharmacokinetics of BMS-753493 in Subjects With Advanced Cancer (Schedule 1)
Brief Title: A Phase 1/2 Study of Epofolate (BMS-753493) in Subjects With Advanced Cancer (Schedule 1)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA190-001
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — BMS-753493

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Epofolate

INTERVENTIONS:
Drug: Epofolate — Intravenous solution, intravenous, initially 3 patients will be treated and if there is a DLT then additional 3 patients will be treated in that dose level. 3-5 minute IV bolus on Days 1, 4, 8 and 11 of a 21-day cycle, until the disease progresses
  Other Names: BMS-753493

SUMMARY:
The purpose of this clinical research study is to study the safety of Epofolate (BMS-753493) in patients with advanced cancers (in Phase 1 portion) and to determine whether Epofolate (BMS-753493) can shrink or slow the growth of the cancer in patients with advanced ovarian, renal or breast cancer (in Phase 2 portion).

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer, excluding cancer in the blood
* Availability of 10 tumor tissue slides

Exclusion:

* Known brain metastases
* Severe nerve damage
* Significant cardiovascular disease
* Inadequate blood counts
* Inadequate liver or kidney function
* Inadequate thyroid function or uncontrolled thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose, the Dose Limiting Toxicity and the recommended dose of Epofolate (BMS-753493) | at the end of the study

SECONDARY OUTCOMES:
To evaluate the safety and exposure levels of Epofolate (BMS-753493) in the body and the anticancer activity of Epofolate (BMS-753493) | every 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (3):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Local Institution, Rotterdam, Netherlands

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx